CLINICAL TRIAL: NCT05965219
Title: A Phase 1, Open-label, Three-Part, Fixed-Sequence Trial in Healthy Adult Participants to Evaluate the Effects of Itraconazole and Carbamazepine on the Single-Dose Pharmacokinetics of Emraclidine, and the Effect of Emraclidine on the Single-Dose Pharmacokinetics of Metformin
Brief Title: A Trial to Evaluate the Effects of Itraconazole and Carbamazepine on the Pharmacokinetics of Emraclidine and of Emraclidine on the Pharmacokinetics of Metformin in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerevel Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CVL-231-HV-1010
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Itraconazole; Carbamazepine; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: Emraclidine Followed by Itraconazole + Emraclidine (Experimental): Participants will receive a single oral dose of emraclidine 10 milligrams (mg) on Day 1 in Treatment Period (TP) 1 followed by itraconazole 200 mg, orally, twice daily (BID) on Day 1 and once daily (QD) from Days 2 to 14, with a single oral dose of emraclidine 10 mg co-administered on Day 5 in TP 2.
  Interventions: Drug: Emraclidine; Drug: Itraconazole
- Part B: Emraclidine Followed by Carbamazepine + Emraclidine (Experimental): Participants will receive a single oral dose of emraclidine 30 mg on Day 1 in TP 1 followed by carbamazepine 100 mg BID from Days 1 to 3, 200 mg BID from Days 4 to 6, and 300 mg BID from Days 7 to 19, orally, with a single oral dose of emraclidine 30 mg on Day 16 in TP 2.
  Interventions: Drug: Emraclidine; Drug: Carbamazepine
- Part C: Metformin Followed by Emraclidine + Metformin (Experimental): Participants will receive a single oral dose of metformin 850 mg on Day 1 in TP 1 followed by emraclidine 30 mg, orally, QD for Days 1 to 10, with a single oral dose of metformin 850 mg co-administered on Day 8 in TP 2.
  Interventions: Drug: Emraclidine; Drug: Metformin

INTERVENTIONS:
Drug: Emraclidine — Emraclidine tablets.
Drug: Itraconazole — Itraconazole oral solution.
  Other Names: Sporanox
  Arms: Part A: Emraclidine Followed by Itraconazole + Emraclidine
Drug: Carbamazepine — Carbamazepine tablets.
  Other Names: Tegretol-XR
  Arms: Part B: Emraclidine Followed by Carbamazepine + Emraclidine
Drug: Metformin — Metformin tablets.
  Other Names: Glucophage
  Arms: Part C: Metformin Followed by Emraclidine + Metformin

SUMMARY:
The primary purpose of the study is to evaluate the effect of itraconazole, a strong cytochrome P450 (CYP) 3A4 inhibitor, on the pharmacokinetics (PK) of emraclidine and metabolite CV-0000364 in Part A, the effect of carbamazepine, a strong CYP3A4 inducer, on the PK of emraclidine and metabolite CV-0000364 in Part B, and to evaluate the effect of emraclidine on the PK of metformin in Part C in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* Healthy as determined by medical evaluation, including medical and psychiatric history, physical and neurological examinations, ECG, vital sign measurements, and laboratory test results, as evaluated by the investigator.
* Body mass index of 18.5 to 35.0 kilograms per square meter (kg/m^2), inclusive, and a total body weight ≥50 kilograms (kg) (110 pounds [lbs]).

Inclusion Criteria for Part A:

* Male and female (women of nonchildbearing potential only) participants, ages 18 to 55 years, inclusive, at the time of signing the informed consent form (ICF).

Inclusion Criteria for Part B:

* Male and female (women of nonchildbearing potential only) participants, ages 18 to 55 years, inclusive, at the time of signing the ICF.

Inclusion Criteria for Part C:

* Male and female (both women of childbearing and nonchildbearing potential) participants, ages 18 to 55 years, inclusive, at the time of signing the ICF.
* Sexually active women of childbearing potential must agree to use at least an acceptable birth control method during the trial and for 7 days after the last dose of IMP. Acceptable birth control methods that result in a failure rate of more than 1% per year include the following:

  * Progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mode of action
  * Male or female condom with or without spermicide
  * Cap, diaphragm, or sponge with spermicide

Exclusion Criteria for All Participants:

* Current or past history of significant cardiovascular, pulmonary, gastrointestinal, renal, hepatic, metabolic, genitourinary, endocrine (including diabetes mellitus, thyroid disorders), malignancy, hematological, immunological, neurological, or psychiatric disease that, in the opinion of the investigator or medical monitor, could compromise either participant safety or the results of the trial.
* "Yes" responses for any of the following items on the C-SSRS (within the individual's lifetime):

  * Suicidal Ideation Item 3 (Active Suicidal Ideation With Any Methods [Not Plan] Without Intent to Act)
  * Suicidal Ideation Item 4 (Active Suicidal Ideation With Some Intent to Act, Without Specific Plan)
  * Suicidal Ideation Item 5 (Active Suicidal Ideation With Specific Plan and Intent)
  * Any of the Suicidal Behavior items (Actual Attempt, Interrupted Attempt, Aborted Attempt, or Preparatory Acts/Behavior)
* "Yes" responses for any of the following items on the C-SSRS (within past 12 months):

  * Suicidal Ideation Item 1 (Wish to be Dead)
  * Suicidal Ideation Item 2 (Non-Specific Active Suicidal Thoughts)
* Serious risk of suicide in the opinion of the investigator is also exclusionary.
* Any condition or surgery that could possibly affect drug absorption, including, but not limited to, bowel resections, bariatric weight loss surgery/procedures, gastrectomy, and cholecystectomy.
* Positive result for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen, hepatitis B total core antibody, or hepatitis C antibody with detectable viral ribonucleic acid (RNA) levels at Screening.
* Positive drug screen (including cotinine and tetrahydrocannabinol [THC]) or a positive test for alcohol.

Exclusion Criteria for Part A:

* History of presence of any of the following and deemed clinically significant by the investigator or designee and confirmed by the medical monitor:

  * Ventricular dysfunction or risk factors for torsades de pointes (e.g., heart failure, cardiomyopathy, family history of long-QT syndrome)
* Any of the following clinical laboratory test results at the Screening Visit or Check-in (Day -1), which can be confirmed by a single repeat measurement, if deemed necessary:

  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > upper limit of normal (ULN).
  * Total bilirubin >ULN. If Gilbert's syndrome is suspected, total bilirubin >ULN is acceptable if the conjugated or direct bilirubin fraction is <20% of total bilirubin.
  * Hypokalemia (potassium levels < lower limit of normal [LLN] millimoles per liter [mmol/L]), and/or hypomagnesemia (magnesium levels <1.2 milligrams per deciliter [mg/dL]; <0.5 mmol/L), and/or hypocalcemia (corrected serum calcium <8.0 mg/dL or ionized calcium <1.0 mmol/L).

Exclusion Criteria for Part B:

* Participants positive for human leukocyte antigen (HLA)-B*1502 or HLA-A*3101.
* Family history of drug reaction with eosinophilia and systemic symptoms (DRESS).
* Family history of porphyria.
* History of cardiac conduction disturbance including second- and third-degree atrioventricular heart block.
* Any of the following clinical laboratory test results at the Screening Visit or Check-in (Day -1), which can be confirmed by a single repeat measurement:

  * Platelets, white blood cell count, absolute neutrophil count, or hemoglobin <LLN.
  * Serum sodium <LLN.
* Any of the following clinical laboratory test results at the Screening Visit or Check-in (Day -1), which can be confirmed by a single repeat measurement, if deemed necessary:

  * AST or ALT >ULN.
  * Total bilirubin >ULN. If Gilbert's syndrome is suspected, total bilirubin >ULN is acceptable if the conjugated or direct bilirubin fraction is <20% of total bilirubin.

Exclusion Criteria for Part C:

* Any of the following clinical laboratory test results at the Screening Visit or Check-in (Day -1), as assessed by the central laboratory and confirmed by a single repeat measurement, if deemed necessary:

  * AST or ALT ≥2 × ULN.
  * Total bilirubin >1.5 × ULN. If Gilbert's syndrome is suspected, total bilirubin >1.5 × ULN is acceptable if the conjugated or direct bilirubin fraction is <20% of total bilirubin.
* Female participants who are pregnant, breastfeeding, or planning to become pregnant during IMP treatment or within 7 days after the last dose of IMP. Women of childbearing potential must have a negative serum pregnancy test result at the Screening Visit and a negative urine pregnancy test result at Check-in.

[Note: Other inclusion and exclusion criteria as per protocol may apply.]

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Part A: Maximum Observed Plasma Concentration (Cmax) of Emraclidine and its Metabolite CV-0000364 | Pre-dose and at multiple time points post-dose from Day 1 in TP 1 up to Day 15 in TP 2 of Part A
Part B: Cmax of Emraclidine and its Metabolite CV-0000364 | Pre-dose and at multiple time points post-dose from Day 1 in TP 1 up to Day 20 in TP 2 of Part B
Part C: Cmax of Metformin | Pre-dose and at multiple time points post-dose from Day 1 in TP 1 up to Day 11 in TP 2 of Part C
Part A: Area Under the Plasma Concentration-time Curve from Time Zero to Last Specified Sampling Time (AUC0-t) of Emraclidine and its Metabolite CV-0000364 | Pre-dose and at multiple time points post-dose from Day 1 in TP 1 up to Day 15 in TP 2 of Part A
Part B: AUC0-t of Emraclidine and its Metabolite CV-0000364 | Pre-dose and at multiple time points post-dose from Day 1 in TP 1 up to Day 20 in TP 2 of Part B
Part C: AUC0-t of Metformin | Pre-dose and at multiple time points post-dose from Day 1 in TP 1 up to Day 11 in TP 2 of Part C
Part A: Area Under the Plasma Concentration-time Curve from Time Zero to Infinity (AUCinf) of Emraclidine and its Metabolite CV-0000364 | Pre-dose and at multiple time points post-dose from Day 1 in TP 1 up to Day 15 in TP 2 of Part A
Part B: AUCinf of Emraclidine and its Metabolite CV-0000364 | Pre-dose and at multiple time points post-dose from Day 1 in TP 1 up to Day 20 in TP 2 of Part B
Part C: AUCinf of Metformin | Pre-dose and at multiple time points post-dose from Day 1 in TP 1 up to Day 11 in TP 2 of Part C

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) Based on Severity | From the first dose up to 1 month following last dose with investigational medicinal product (IMP) in each part of the study
Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Values | Up to end of treatment in each part of the study (up to an average of 15 days)
Number of Participants With Clinically Significant Changes in Vital Sign Measurements | Up to end of treatment in each part of the study (up to an average of 15 days)
Number of Participants With Clinically Significant Changes in Laboratory Assessments | Up to end of treatment in each part of the study (up to an average of 15 days)
Number of Participants With Clinically Significant Changes in Physical and Neurological Examination Results | Up to end of treatment in each part of the study (up to an average of 15 days)
Changes in Suicidality Assessed Using the Columbia Suicide Severity Rating Scale (C-SSRS) Score | Up to end of treatment in each part of the study (up to an average of 15 days)
  The C-SSRS includes 'yes' or 'no' responses for assessment of suicidal ideation and behavior as well as numeric ratings for the severity of ideation, if present (from 1 to 5, with 5 being the most severe). Greater lethality or potential lethality of suicidal behaviors (endorsed on the behavior subscale) indicates increased risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Overland Park, Kansas, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No